CLINICAL TRIAL: NCT02373891
Title: Study to Evaluate the Effect of Food on the Pharmacokinetics of Surfolase CR Tablet in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hyundai Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HT-002-04
Record Dates: First submitted 2015-02-11; First posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- T1 (Experimental)
  Interventions: Drug: Surfolase CR
- T0 (Experimental)
  Interventions: Drug: Surfolase CR

INTERVENTIONS:
Drug: Surfolase CR — T1: Surfolase CR (Acebrophylline 200mg) administration after fat intake Surfolase CR(Acebrophylline 200mg) administrated fasting or fat intake at D1 and D8 a.m. 8:00
  Arms: T1
Drug: Surfolase CR — T0: Surfolase CR(Acebrophylline 200mg) fasting administration Surfolase CR(Acebrophylline 200mg) administrated fasting or fat intake at D1 and D8 a.m. 8:00
  Arms: T0

SUMMARY:
Acebrophylline is metabolized by being separated into Ambroxol and 7-theophylline when orally administered as a salt composed of an acid-base as a compound that was synthesized by and chloride (salifying) the ambroxol to 7-theophylline. Acebrophylline is selectively applied to the bronchial or lung tissue and inhibit the activity of phospholipase bronchoalveolar shows the expectorant action to raise the surface activity of the alveolar, leukotrienes (LTs) and by suppressing the production of prostaglandins (PGs), showed potent anti-inflammatory activity, bronchial was celebrated by reducing the bronchial hyperreactivity to normal state is allowed to recuperate or extended.

It was developed to improve compliance improve pharmaceutically Acebrophylline that intake twice daily 100mg to Surfolase CR that intake once daily 200mg

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between the ages of 20 and 55 years, BMI >18.5, <25, inclusive

   *Body mass index(kg/m2) = weight(kg)/(height(m)2)
2. Subject who don't have congenital or chronic diseases and have no abnormal medical examination results.
3. Subject is healthy (no clinically relevant findings in any of the investigations of the pre-examination) as judged by the investigator

   * Hematology tests: WBC with differential count, RBC, Hemoglobin, Hematocrit, Platelet, PT(INR)/aPTT
   * Blood chemistry tests: Calcium, Inorganic Phosphate, Fasting Glucose, BUN, Creatinine, Cholesterol, Total Protein, Albumin, Total Bilirubin, Alkaline phosphatase, AST, ALT, r-GT, LDH, TG, K, Na, Cl, uric acid, CPK
   * Immune serum tests: HBsAg, anti-HCV Ab, anti-HIV Ag/Ab, β-hCG
   * Urinalysis: Specific Gravity, pH, Protein, Glucose, Ketone, RBC, Urobilinogen, Bilirubin, Nitrite, WBC, Color, Turbidity, Sediment, Microscopy
   * Urine drug screening tests: Amphetamine, Barbiturate, Morphine, Benzodiazepine, Cocaine 4) If you are a woman, you must be a negative pregnancy test at screening.
   * Postmenopausal (no period for at least two years)
   * Surgical sterilization (Hysterectomy or bilateral oophorectomy, tubal ligation)
   * Before the screening, interfile male partner and this man is the sole partner of that person
   * Before Investigational product first dose administered at least 14 days before the start appropriate contraception until at least 28 days.

     5) If you are a male and sexually active women of childbearing age, during the trial period contraception (condoms, etc.) and clinical trial duration, and IND maintaining adequate contraception up to 28 days after the last dose, and one party must agree that you will not donate sperm 6) Subjects who signed and dated in informed consent form indicating that the subject has decided to participate in the study after being informed of all pertinent aspects of the study

Exclusion Criteria:

1. Subject with known for hypersensitivity reaction to acebrophylline, xanthine and food.
2. Patients with genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
3. Subject with serious active cardiovascular, respiratory, hepatologic, renal, hematologic, gastrointestinal, immunologic, dermal, neurologic, or psychological disease or history of such disease
4. Subject with known for history of gastrointestinal disease or gastrointestinal surgery which affect on the absorption drug
5. Subjects with any of the following condition in screening (blood pressure, 12-lead ECG, blood, urinalysis, etc.)
6. Subject with any of the following conditions in laboratory test

   * AST or ALT > Upper normal limit × 1.25
   * Total bilirubin > Upper normal limit × 1.5
7. If the estimated GFR < 80mL/min/1.73m2 using MDRD formula.

   ※ MDRD equation (mL/min/1.73m2)

   : GFR = 175 x Scr-1.154 x age-0.203
8. Systolic blood pressure <=90mmHg or diastolic blood pressure >=150mmHg or a person showing the corresponding figures <=50mmHg or >=100mmHg in vital signs.
9. Who has history of drug abuse (especially hypnotic, central acting analgesics, psychotropic drugs, such as opiates or central nervous system acting drug) or shows positive reactions to drug of abuse in urine drug screening tests.
10. Excessive caffeine and alcohol intake, smoking person(caffeine: > 5cups/day, alcohol: >210g/week, tobacco: > 10 cagarettes/day)
11. Person cannot be non-smoking, non-alcohol during the hospital stay.
12. Use of any prescription medication within 14 days prior to study medication dosing or use of any medication such as over-the-counter medication including oriental medication within 7 days prior to study medication dosing
13. Participation in any clinical investigation within 60days prior to study medication dosing
14. Subjects with whole blood donation within 60days, component blood donation within 30days
15. Women who are pregnant or breast-feeding
16. Person who cannot eat, including high-fat diet (more than 900kcal, containing more that 35% fat) that served during the trial period
17. Person can not prohibit the consumption of grapefruit-containing food during the trial period.
18. Subjects with decision of nonparticipation through investigator's review due to laboratory test results or other excuse such as non-responding to request or instruction by investigator

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Ambroxol AUClast, Cmax | Fasting medication: 0 h (before intake), 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 14, 24, 36 h (17 times), Fat meal medication: 0 h (before intake), 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 14, 24, 36h
Ambroxol AUCinf, Tmax, t1/2 | Fasting medication: 0 h (before intake), 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 14, 24, 36 h (17 times), Fat meal medication: 0 h (before intake), 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 14, 24, 36h

CONTACTS AND LOCATIONS:
Overall Officials: Park, Principal Investigator — Severance Hospital